CLINICAL TRIAL: NCT06126874
Title: Additional Effects of Aerobic and Resistance Exercise Training to Pelvic Floor Muscle Training in Urinary Incontinence and Erectile Dysfunction After Radical Prostatectomy
Brief Title: Additional Effects of Aerobic and Resistance Exercises to Pelvic Floor Muscle Training After Radical Prostatectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SERAP ÖZGÜL, Prof. Dr., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA-23054
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Incontinence; Erectile Dysfunction Following Radical Prostatectomy
Keywords: men's health; radical prostatectomy; urinary incontinence; erectile dysfunction; pelvic floor muscle training; aerobic exercise; resistance exercise; Kegel exercise
MeSH Terms: conditions — Urinary Incontinence; Erectile Dysfunction | interventions — Patient Education as Topic; Resistance Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient education, Pelvic floor muscle training, Aerobic and Resistance exercise trainings (Experimental): Patient Education: Individuals in both study groups will be provided with patient education through verbal and visual presentations.
  Pelvic Floor Muscle Training (PFMT): In PFMT, voluntary maximal and submaximal contractions for strength and endurance training of pelvic floor muscles will be taught and individuals will continue PFMT as a home exercise program.
  Aerobic Exercise Training: Aerobic exercise training will be planned 3 days a week, 1 day on the routine clinic day with a treadmill ergometer and 2 days as a home program in the form of brisk walking outside the clinic (e.g. outdoors or in a suitable environment).
  Resistance Exercise Training: Resisted exercise training will be planned 2 days a week, 1 day in the clinic and 1 day outside the clinic as a home program, and 12 different exercises for large muscle groups with dumbbells and weight sets, resistance bands (therabands) will be used in the training.
  Interventions: Other: Patient Education; Other: Pelvic Floor Muscle Training; Other: Aerobic Exercise Training; Other: Resistance Exercise Training
- Patient education and Pelvic floor muscle training (Active Comparator): Patient Education: Individuals in both study groups will be provided with patient education through verbal and visual presentations.
  Pelvic Floor Muscle Training (PFMT): In PFMT, voluntary maximal and submaximal contractions for strength and endurance training of pelvic floor muscles will be taught and individuals will continue PFMT as a home exercise program.
  Interventions: Other: Patient Education; Other: Pelvic Floor Muscle Training

INTERVENTIONS:
Other: Patient Education — Individuals in both study groups will be provided with patient education through verbal and visual presentations. In the content of patient education; information about the importance of the research topic and the content of the study through anatomical models and short animations, lifestyle recommendations for urinary incontinence symptoms (avoiding bladder irritants such as alcohol, caffeine, tea, spicy foods, acidic foods and chocolate, regulating water / fluid consumption, recommendations for attention to bowel regularity and increasing physical activity levels) and recommendations for sexual functioning (coitus positions that facilitate erection, recommendations for reshaping the sexual schema, recommendations for the physical dimension of sexual health) will be given.
Other: Pelvic Floor Muscle Training — In PFMT, voluntary maximal and submaximal contractions for strength and endurance training of pelvic floor muscles will be taught and individuals will continue PFMT as a home exercise program. In the first 2 weeks of PFMT, individuals will perform 3 sessions of exercise per day. In each 2-week control, the number of sessions will be increased by 1 session and PFMT application will be completed with 5 sessions per day in the study.
Other: Aerobic Exercise Training — Aerobic exercise training will be planned 3 days a week, 1 day on the routine clinic day with a treadmill ergometer and 2 days as a home program in the form of brisk walking outside the clinic (e.g. outdoors or in a suitable environment).The intensity of aerobic exercise training will be planned according to the Maximal Heart Rate (MHR) method and Modified Borg Scale (MBS). In the first 2 weeks in the clinic, training will be started with 50 min (+10 min warm-up and cool-down) at 60% of the MHR, the exercise intensity will be increased by 5% every 2 weeks, and the program will be terminated by providing exercise training at 85% of the MHR in the 10th-12th week. Patients will be asked to adjust the intensity of aerobic exercise outside the clinic to correspond to the 12-14 (slightly difficult) degree of perceived fatigue according to the MBS.
  Arms: Patient education, Pelvic floor muscle training, Aerobic and Resistance exercise trainings
Other: Resistance Exercise Training — Resisted exercise training will be planned 2 days a week, 1 day in the clinic and 1 day outside the clinic as a home program, and 12 different exercises for large muscle groups with dumbbells and weight sets, resistance bands (therabands) will be used in the training. These exercises are leg press, leg extension, leg curl, squat, seated row, lateral pull down, biceps curl, triceps extension, dumble fly, lateral raises, bench press and abdominal crunch. Exercises will be performed with free weights (dumbbells), resistance bands (therabands) or body weight.
  Arms: Patient education, Pelvic floor muscle training, Aerobic and Resistance exercise trainings

SUMMARY:
In the literature, studies about urinary symptoms after radical prostatectomy (RP) are generally focused on urinary incontinence (UI), and studies about sexual symptoms are focused on erectile dysfunction (ED). In the management of these symptoms, the effects of pharmacological agents (duloxetine/antimuscarinics and PDE5-I) and/or local approaches (pelvic floor muscle training-PFMT, vacuum erection devices) have been emphasized. In these studies, the results are contradictory and the level of evidence is low. The effects of aerobic and resistance exercise training on urinary, sexual and general health after RP have not been revealed from a holistic and multidisciplinary perspective. Therefore, the aim of this study was to investigate the additional effects of aerobic and resistance exercise trainings to pelvic floor muscle training on urinary incontinence and erectile dysfunction after radical prostatectomy in a randomized controlled design.

The study will include volunteers aged 40 years and older (Mini Mental test score of 24 and above for individuals aged 65 years and older) with symptoms of UI and/or ED after RP. The study is designed as a randomized controlled trial. Individuals who meet the inclusion criteria and agree to participate in the study will be randomly assigned to 2 separate groups. Subjects in the research group will receive patient education, PFMT, and aerobic and resistance exercise trainings; subjects in the control group will receive only patient education and PFMT. The study period is 12 weeks. Individuals will be evaluated at 2 separate time periods, at the beginning of the study and at the end of the 12th week.

DETAILED DESCRIPTION:
In the literature, studies about urinary symptoms after radical prostatectomy (RP) are generally focused on urinary incontinence (UI), and studies about sexual symptoms are focused on erectile dysfunction (ED). In the management of these symptoms, the effects of pharmacological agents (duloxetine/antimuscarinics and PDE5-I) and/or local approaches (pelvic floor muscle training-PFMT, vacuum erection devices) have been emphasized. In these studies, the results are contradictory and the level of evidence is low. The effects of aerobic and resistance exercise training on urinary, sexual and general health after RP have not been revealed from a holistic and multidisciplinary perspective. Therefore, the aim of this study was to investigate the additional effects of aerobic and resistance exercise trainings to pelvic floor muscle training on urinary incontinence and erectile dysfunction after radical prostatectomy in a randomized controlled design.The hypotheses of the study are as follows:

* H1: After radical prostatectomy, aerobic and resistance exercise trainings in addition to pelvic floor muscle training (PFMT) provides greater improvement in objective UI severity, urinary symptoms and incontinence-specific quality of life.
* H2: After radical prostatectomy, aerobic and resistance exercise trainings in addition to PFMT provides greater improvement in in penile length.
* H3: After radical prostatectomy, aerobic and resistance exercise trainings in addition to PFMT provides greater improvement in erectile function and sexual health.
* H4: After radical prostatectomy, aerobic and resistance exercise trainings in addition to PFMT provides greater improvement in peripheral muscle strength.
* H5: After radical prostatectomy, aerobic and resistance exercise trainings in addition to PFMT provides greater improvement in functional exercise capacity.
* H6: After radical prostatectomy, aerobic and resistance exercise trainings in addition to PFMT provides greater improvement in general health and quality of life.

The study will include volunteers aged 40 years and older (Mini Mental test score of 24 and above for individuals aged 65 years and older) with symptoms of UI and/or ED after RP. The study is designed as a randomized controlled trial. Individuals who meet the inclusion criteria and agree to participate in the study will be randomly assigned to 2 separate groups. Subjects in the research group will receive patient education, PFMT, and aerobic and resistance exercise trainings; subjects in the control group will receive only patient education and PFMT. The study period is 12 weeks. Individuals will be evaluated at 2 separate time periods, at the beginning of the study and at the end of the 12th week. Subjective severity of incontinence and its impact on life will be assessed with the International Consultation Incontinence Questionnaire-Short Form (ICIQ-SF). The International Consultation on Incontinence Questionnaire-Male Lower Urinary Tract Symptoms (ICIQ-MLUTS) scale will be used to question the severity of lower urinary tract symptoms. Erectile function and sexual function will be questioned with the International Erectile Function Form -15 (IIEF-15). Depression Anxiety Stress Scale-21 (DASS-21) will be used to evaluate the depression, anxiety and stress levels of the patients. The World Health Organization Quality of Life Questionnaire-Short Form (WHOQOL-BREF) will be used to question the general quality of life of the individuals. Objective severity of incontinence will be evaluated with a 1-hour pad test. Peripheral muscle strength will be evaluated with a hand-held dynamometer and functional exercise capacity of the individuals will be evaluated by 6-Minute Walking Test (6-MWT).

ELIGIBILITY:
Inclusion Criteria:

* Individuals with localized prostate cancer (Stage I-II) undergoing Robot-Assisted Laparoscopic or Open Bilateral Nerve-Sparing Radical Prostatectomy
* being married or having a partner
* lack of cooperation problems with the assessments and interventions in the study
* Being 40 years or older

Exclusion Criteria:

* Acute disease status (e.g. urinary tract infection, respiratory infection, presence of interstitial cystitis, bladder or gastrointestinal bleeding),
* Acute surgical condition (within the first 3 weeks after prostatectomy),
* Presence of neurological disease or neurogenic bladder,
* Preoperative incontinence,
* Bladder or other prostate surgery prior to prostatectomy,
* Preoperative/postoperative pelvic radiotherapy,
* Reporting preoperative ED or sexual dysfunction other than ED,
* Have any medical condition that may limit their exercise training,
* Individuals over 65 years of age with a Mini Mental Test score of less than 24 (a score of less than 24 indicates mild/moderate dementia)

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
International Consultation on Incontinence Questionnaire- Short Form (ICIQ-SF) Score | Change in severity of incontinence from baseline to the end of the 12th week.
  The ICIQ-UI Short Form is a questionnaire for evaluating the frequency, severity and impact of urinary incontinence on quality of life (QoL) in men and women in research and clinical practice.
International Index of Erectil Function-15 ( IIEF-15) Score | Change in severity of erectile function from baseline to the end of the 12th week.
  The IIEF-15 is a multidimensional scale that can be used to evaluate ED. It has five subdomains: Erectile Function ( items 1,2,3,4,5,15), Orgasmic Function ( items 9,10), Sexual Desire (items 11,12), Intercourse Satisfaction ( items 6,7,8), Overall Satisfaction (items 13,14).

SECONDARY OUTCOMES:
1-hour Pad Test Score | Change in severity of incontinence from baseline to the end of the 12th week.
  1-Hour Pad test is a non-invasive test that is widely used in the evaluation of objective UI severity.
Penile Length | Change in penile length from baseline to the end of the 12th week.
  Penile length will be measured by the therapist with the help of a ruler. This is a non-invasive objective measurement method used in the literature to measure the penile length of individuals after prostatectomy.
Peripheral Muscle Strength | Change in strength of peripheral muscles from baseline to the end of the 12th week.
  Peripheral muscle strength will be evaluated with a hand-held dynamometer. The handheld dynamometer is a non-invasive and routinely used objective assessment tool preferred in the clinic for strength measurement. Studies have shown that handheld digital dynamometers are useful tools to objectively assess muscle strength before and after intervention and to demonstrate the effectiveness of treatment. In our study, within the scope of peripheral muscle strength measurement, static strength measurements will be performed in shoulder flexion-extension, shoulder abduction-adduction, elbow flexion-extension, hip flexion-extension, knee flexion-extension, and ankle dorsal and plantar flexion.
Functional Exercise Capacity | Change in distance from baseline to the end of the 12th week.
  Functional exercise capacity of individuals will be evaluated with the 6 Minute Walking Test (6MWT). The 6MWT is a simple and non-invasive test that evaluates the submaximal functional exercise capacity of individuals in 6 minutes on a hard and flat surface, does not require special equipment or advanced training, and has been shown to be reliable and valid in various patient populations in the literature.
International Consultation On Incontinence- Male Lower Urinary Tract Symptoms (ICIQ-MLUTS) Score | Change in lower urinary system symptoms scores from baseline to the end of the 12th week.
  The ICIQ-MLUTS is a questionnaire for evaluating male lower urinary tract symptoms and impact on quality of life (QoL) in research and clinical practice. It has four subdomains: Voiding Score (2-6 items), Incontinence Score (7-12 items), Frequency of urination during the day (13th item), Frequency of urination during the night (14th item)
Depression Anxiety and Stress Scale-21 (DASS-21) Score | Change in level of depression, anxiety and stress level from baseline to the end of the 12th week.
  The DASS-21 is a self-report scale designed to measure the negative emotional states of depression, anxiety and stress. It contains 21 questions totally and 7 questions for each symptoms. Depression: dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest / involvement, anhedonia and inertia. (Items 3, 5, 10, 13, 16, 17, 21). Anxiety: autonomic arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect. (Items 2, 4, 7, 9, 15, 19, 20). Stress: levels of chronic nonspecific arousal, difficulty relaxing, nervous arousal, and being easily upset / agitated, irritable / over-reactive and impatient (Items 1, 6, 8, 11, 12, 14, 18).
World Health Organization Quality of Life Brief Version (WHOQOL-BREF) Score | Change in quality of life from baseline to the end of the 12th week.
  The World Health Organization Quality of Life Scale-Short Form (WHOQOL-BREF) will be used to question the general quality of life of individuals.The WHOQOL-BREF addresses four quality of life domains: physical health, psychological health, social relationships and environment.

CONTACTS AND LOCATIONS:
Overall Officials: Serap ÖZGÜL, Prof, Principal Investigator — Hacettepe University, Department of Physiotherapy and Rehabilitation; Naşide MANGIR, Assoc Prof, Study Director — Hacettepe University, Department of Urology
Locations (1):
- Mustafa Enis Dilekmen, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Avery K, Donovan J, Peters TJ, Shaw C, Gotoh M, Abrams P. ICIQ: a brief and robust measure for evaluating the symptoms and impact of urinary incontinence. Neurourol Urodyn. 2004;23(4):322-30. doi: 10.1002/nau.20041. PMID 15227649
- [Background] Neijenhuijs KI, Holtmaat K, Aaronson NK, Holzner B, Terwee CB, Cuijpers P, Verdonck-de Leeuw IM. The International Index of Erectile Function (IIEF)-A Systematic Review of Measurement Properties. J Sex Med. 2019 Jul;16(7):1078-1091. doi: 10.1016/j.jsxm.2019.04.010. Epub 2019 May 27. PMID 31147249
- [Background] Jorgensen L, Lose G, Andersen JT. One-hour pad-weighing test for objective assessment of female urinary incontinence. Obstet Gynecol. 1987 Jan;69(1):39-42. PMID 3796918
- [Background] Greenstein A, Dekalo S, Chen J. Penile size in adult men-recommendations for clinical and research measurements. Int J Impot Res. 2020 Mar;32(2):153-158. doi: 10.1038/s41443-019-0157-4. Epub 2019 Jun 6. PMID 31171853
- [Background] Kwon YS, Farber N, Yu JW, Rhee K, Han C, Ney P, Hong JH, Lee P, Gupta N, Kim WJ, Kim IY. Longitudinal recovery patterns of penile length and the underexplored benefit of long-term phosphodiesterase-5 inhibitor use after radical prostatectomy. BMC Urol. 2018 May 9;18(1):37. doi: 10.1186/s12894-018-0341-8. PMID 29739455
- [Background] Chamorro C, Armijo-Olivo S, De la Fuente C, Fuentes J, Javier Chirosa L. Absolute Reliability and Concurrent Validity of Hand Held Dynamometry and Isokinetic Dynamometry in the Hip, Knee and Ankle Joint: Systematic Review and Meta-analysis. Open Med (Wars). 2017 Oct 17;12:359-375. doi: 10.1515/med-2017-0052. eCollection 2017. PMID 29071305
- [Background] Chamorro C, Arancibia M, Trigo B, Arias-Poblete L, Jerez-Mayorga D. Absolute Reliability and Concurrent Validity of Hand-Held Dynamometry in Shoulder Rotator Strength Assessment: Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2021 Sep 3;18(17):9293. doi: 10.3390/ijerph18179293. PMID 34501883
- [Background] Mertoglu O, Ucer O, Ceylan Y, Bozkurt O, Gunlusoy B, Albaz AC, Demir O; Aegean Study Group of Society of Urological Surgery. Reliability and Validity of the Turkish Language Version of the International Consultation on Incontinence Questionnaire - Male Lower Urinary Tract Symptoms. Int Neurourol J. 2016 Jun;20(2):159-63. doi: 10.5213/inj.1630460.230. Epub 2016 Jun 24. PMID 27377949
- [Background] Henry JD, Crawford JR. The short-form version of the Depression Anxiety Stress Scales (DASS-21): construct validity and normative data in a large non-clinical sample. Br J Clin Psychol. 2005 Jun;44(Pt 2):227-39. doi: 10.1348/014466505X29657. PMID 16004657
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712
- [Background] Giannitsi S, Bougiakli M, Bechlioulis A, Kotsia A, Michalis LK, Naka KK. 6-minute walking test: a useful tool in the management of heart failure patients. Ther Adv Cardiovasc Dis. 2019 Jan-Dec;13:1753944719870084. doi: 10.1177/1753944719870084. PMID 31441375
- [Background] Bellet RN, Adams L, Morris NR. The 6-minute walk test in outpatient cardiac rehabilitation: validity, reliability and responsiveness--a systematic review. Physiotherapy. 2012 Dec;98(4):277-86. doi: 10.1016/j.physio.2011.11.003. Epub 2012 May 16. PMID 23122432
- [Background] Rasekaba T, Lee AL, Naughton MT, Williams TJ, Holland AE. The six-minute walk test: a useful metric for the cardiopulmonary patient. Intern Med J. 2009 Aug;39(8):495-501. doi: 10.1111/j.1445-5994.2008.01880.x. PMID 19732197